CLINICAL TRIAL: NCT04710914
Title: Comparison of Extubation Delay After Prolonged Sedation With Inhaled Isoflurane Using the MIRUS® Device or Continuous Intravenous Midazolam in Patients With Septic Shock in Intensive Care
Brief Title: Comparison of Extubation Delay After Prolonged Sedation
Acronym: ISOREA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID epidemic and sedation practices that have completely changed: the standard sedative is now propofol rather than midazolam.
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/0348/HP
Record Dates: First submitted 2020-12-29; First posted 2021-01-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Isoflurane; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sedation by inhaled isoflurane (Experimental): sedation by midazolam with the MIRUS device
  Interventions: Drug: Prolonged sedation with isoflurane
- sedation with intravenous midazolam (Active Comparator): continuation of sedation with intravenous midazolam
  Interventions: Drug: Prolonged sedation with midazolam

INTERVENTIONS:
Drug: Prolonged sedation with isoflurane — Adult patients admitted to the surgical intensive care unit at the Rouen University Hospital for septic shock and requiring sedation for more than 3 days and a maximum of 10 days will be randomised in two groups.
  The experimental group will receive sedation by inhaled isoflurane The control group will receive sedation by intravenous midazolam
  Arms: sedation by inhaled isoflurane
Drug: Prolonged sedation with midazolam — Adult patients admitted to the surgical intensive care unit at the Rouen University Hospital for septic shock and requiring sedation for more than 3 days and a maximum of 10 days will be randomised in two groups.
  The experimental group will receive sedation by inhaled isoflurane The control group will receive sedation by intravenous midazolam
  Arms: sedation with intravenous midazolam

SUMMARY:
This monocentric, prospective, controlled, randomized, single-blind study will be conducted in surgical resuscitation at the Rouen University Hospital. The aim of our research project is to evaluate the extubation time after sedation with inhaled isoflurane compared to conventional intravenous sedation with midazolam, in patients who require prolonged sedation (3 to 28 days) in a context of septic shock. This population is particularly at risk of hypnotic accumulation due to the prolonged duration of use and the increased risk of developing renal or hepatic impairment in connection with septic shock.

Based on data from the literature on shorter durations of up to 96 hours of sedation, the investigators expect a decrease in the time to extubation in patients sedated with isoflurane as well as a better quality of awakening with a decrease in resuscitation delirium. This shortened duration of mechanical ventilation could have beneficial effects on the morbidity associated with prolonged sedation and ventilation: reduction of pneumopathies acquired under mechanical ventilation, reduction of the length of stay in resuscitation and hospitalization.

DETAILED DESCRIPTION:
In intensive care, sedation of patients is frequently used for their management. Combined with analgesia, it provides the comfort essential for the implementation of certain therapies such as mechanical ventilation.

Classically, sedation is based on the combination of a hypnotic and an injectable morphine, most often midazolam and sufentanil. Midazolam is a benzodiazepine with many advantages: few hemodynamic effects, no limited duration of use and good workability. However, its use presents several difficulties in resuscitation:

1. Some patients have accelerated metabolism and resistance to benzodiazepines, either through chronic use of psychotropic or narcotic drugs. These patients develop tolerance phenomena due to enzyme induction. This tachyphylaxis leads to an increased need for midazolam to achieve the therapeutic goal.
2. Some pathologies, such as ARDS, require deep sedation in the initial phase, which may last several days. After this phase, prolonged sedation may be necessary before achieving sufficient improvement to allow sedation to be stopped.
3. The metabolism of midazolam is dependent on liver function and its elimination from renal function. Alteration of these functions, common in resuscitation, results in impaired elimination with accumulation of midazolam and 2 active metabolites, 1-hydroxy-midazolam and 1-hydroxy-midazolam-glucuronide.

These three difficulties may lead to an undesirable prolongation of the sedation period beyond the cessation of midazolam infusion, which is associated with an increase in morbidity such as neuromyopathies, ventilator-associated pneumopathies (VAPP), deliriums and withdrawal syndromes. These complications increase the length of stay and mortality in intensive care units.

For 30 years there has been a growing interest in the use of sedation in resuscitation with volatile halogenated agents (VHAs). These agents, administered by inhalation, have many advantages: short onset of action, good workability, effect not dependent on renal or hepatic function, almost exclusive and predictable respiratory elimination, absence of tachyphylaxis and metabolism not sensitive to enzyme induction. For these reasons, AVHs are widely used in anesthesia in the operating room. The hypnotic action of HVAs is closely correlated with the expired fraction of HVAs. Measured by gas analysers, it allows precise monitoring of the therapeutic effect. In contrast to resuscitation ventilators, all anesthesia ventilators are equipped with evaporation tanks and administration circuits, gas analyzers and associated facilities for their disposal. These technical constraints mean that, despite their many theoretical advantages, AVHs have not been used in resuscitation area.

In the early 2000s, a new device made it possible to use AVH in intensive care: the AnaConDa® system. It made it possible to administer AVH using an evaporator inserted into the patient circuit at the intubation catheter, completely independent of the ventilator. However, this device had several shortcomings in terms of user safety and cost due to the short service life of the consumables.

Since 2016, a new device is available in France: the MIRUS® (Pall Medical, Dreieich, Germany). It has several advantages over AnaConDa® :

* It is equipped with an integrated gas analyzer that allows the automatic adjustment of the AVH flow rate for a concentration target (FeAVH target). This results in greater safety and AVH savings,
* For each AVH with an MA (isoflurane, sevoflurane or desflurane), there is a MIRUS controller with a tank model with a coding and color-coding system to avoid medication errors,
* Filters and reflectors can be used for several days, thus reducing the cost of use.

Among the recent AVHs and as for its use in anesthesia, isoflurane has shown a safety of use in resuscitation on longer uses up to 96 hours without side effects. A recent retrospective study showed no excess mortality after prolonged use of isoflurane (minimum 96 hours, average 506 hours) in post-operative, mainly digestive surgery in patients with sepsis with an average age of 71 years. After medium-length sedation (average duration 52 hours, maximum 96 hours), the recovery and extubation times are shorter than with intravenous sedation with midazolam: 10 minutes versus 250 minutes for the extubation time, but with significant differences in sedation and analgesia protocol compared to our practices. The AVHs have moreover been included in the German recommendations on sedation in resuscitation.

This monocentric, prospective, controlled, randomized, single-blind study will be conducted in surgical resuscitation at the Rouen University Hospital. The aim of our research project is to evaluate the time to extubation after sedation with inhaled isoflurane compared to conventional intravenous sedation with midazolam, in patients requiring prolonged sedation (3 to 28 days) in a context of septic shock. This population is particularly at risk of hypnotic accumulation due to the prolonged duration of use and the increased risk of developing renal or hepatic impairment in connection with septic shock.

Based on data from the literature on shorter durations of up to 96 hours of sedation, the investigators expect a decrease in the time to extubation in patients sedated with isoflurane as well as a better quality of awakening with a decrease in resuscitation delirium. This shortened duration of mechanical ventilation could have beneficial effects on the morbidity associated with prolonged sedation and ventilation: reduction of pneumopathies acquired under mechanical ventilation, reduction of the length of stay in resuscitation and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Major patients,
* Sedated with midazolam and sufentanil for a maximum of 3 days and ventilated invasively,
* Presenting a duration of sedation and invasive ventilation expected after inclusion between 3 days and 10 days,
* Presenting septic shock according to the SEPSIS-3 definition with the following 4 criteria :

  * Clinical suspicion of infection or positive microbiological sample if applicable,
  * Organ Failure: SOFA (Sepsis-related Organ Failure Assessment) ≥ 2 (Annex n°5),
  * Need for vasoactive amines to maintain sufficient organ perfusion pressure,
  * Arterial lactate > 2mmol/l,
* Stabilized septic shock without the need to increase noradrenaline doses over the last 6 hours,
* For women, absence of current pregnancy: negative pregnancy test,
* Subjects affiliated to a social security system.
* If the patient is unable to sign the consent (emergency situation) the consent will be signed by his or her representative ((1) the trusted person, or failing that, (2) a family member, or (3) a relative of the person concerned). In this case, the patient will subsequently be asked for consent to continue the study.

Exclusion Criteria:

* Refusal of the patient to continue the study after waking up,
* Duration of sedation after randomization less than 3 days or more than 10 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
The delay between the first sedation stop and extubation | 10 days
  The delay between the first sedation stop and extubation. This time will be measured from the first interruption of sedation to the patient's extubation. If the patient needs to be resedated prior to extubation, the stop of sedation for the primary endpoint measurement will be the first stop of sedation.

SECONDARY OUTCOMES:
Wake-up time | 10 days
  Measurement of the wake-up time defined by the time between stopping sedation and obtaining a RASS (Richmond Agitation and Sedation Scale) sedation level equal to 0%
Total duration of sedation and mechanical ventilation | 90 days
  Total duration of sedation and mechanical ventilation: data obtained by the ICCA information system (IntelliSpace Critical Care and Anesthesia, Philips) allowing prescription and monitoring in surgical resuscitation.
Total duration of intensive care and hospital stay | 90 days
  Total duration of intensive care and hospital stay: collection of hospitalization records
A measure of overall survival at 90 days defined by the duration between the inclusion date and the date of death. | 90 days
  A measure of overall survival at 90 days defined by the duration between the inclusion date and the date of death. Use of the CDP2 software to consult hospitalization reports and telephone calls from the patient or his or her family in the event of missing data.
Measurement of wake-up time defined by the duration between the day of the first sedation stop and a RASS score of 0, | 10 days
  duration between the day of the first sedation stop and a RASS score of 0between the day of the first sedation stop and a RASS score of 0,
Security | 90 days
  Collection of intercurrent events
Doses of vasopressor, hypnotic and morphine amines administrated | 3 days
  These data are available in the computerized prescriptions. The doses of hypnotics over the entire sedation period will be retrieved in the prescriptions for the midazolam group and extracted from the MIRUS controller using software provided by the manufacturer for the isoflurane group.
Measurement of the number of days without mechanical ventilation | 90 days
  Measurement of the number of days without mechanical ventilation
Measurement of midazolam and 2 active metabolites, 1-OHM and 1-OHMG | 24, 48 and 96 hours
  Quantitative blood assays of midazolam and 2 active metabolites, 1-OHM and 1-OHMG, performed for all patients at randomization, at sedation cessation and after sedation cessation.
Costs of sedative treatments (midazolam and isoflurane) and the devices needed to administer them (syringes and tubing for midazolam, reflector and filter exchanger for isoflurane) | 90 days
  Costs of sedative treatments (midazolam and isoflurane) and the devices needed to administer them (syringes and tubing for midazolam, reflector and filter exchanger for isoflurane)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LEFEVRE-SCELLES, Doctor, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France